CLINICAL TRIAL: NCT03816930
Title: Evaluation of Gingival Health Parameters in Hybrid CAD / CAM Crowns Produced After Different Retraction Processes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Beyza Ünalan Değirmenci, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 05
Record Dates: First submitted 2019-01-17; First posted 2019-01-25 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Periodontal Disease; Gingival Disease
Keywords: CAD/CAM; Gingival retraction
MeSH Terms: conditions — Periodontal Diseases; Gingival Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Mechanical cord usage (Active Comparator): Mechanical retraction
  Interventions: Procedure: mechanical cord usage
- Chemical contained retraction usage (Active Comparator): Chemical retraction
  Interventions: Procedure: mechanical cord usage
- MZ-6 laser tip used throughing (Active Comparator): Laser retraction
  Interventions: Procedure: mechanical cord usage

INTERVENTIONS:
Procedure: mechanical cord usage — Due to the retraction procedures, same preparation conditions will be obtained.
  Other Names: Chemical contained retraction usage; MZ-6 laser tip used throughing

SUMMARY:
Clinically, the gingival retraction dentistry itself has found wide uses. It has achieved the use of subgingival and gingival crowns in fixed prostheses, cervical abrasion in restorative dentistry, management of root caries and root sensitivity, and recently in the use of appropriate measurements to improve the marginal fit of implant prostheses.There are three different retraction procedures described in the literature: mechanical, mechanical-chemical (chemically impregnated cords or matrix in injectable form) and surgery (electrosurgical, laser, cauterization, etc.)The mechanical method of retraction cords is not always suitable for patients' existing pocket depth, the necessity of using different combinations in shallow or deep pockets, the potential for limited bleeding control in chemically impregnated cords and the toxicity values in those who interact with chemical have led researchers to search for alternative methods. Especially inflammed gingiva is very sensitive to mechanical and chemical trauma. Studies have reported that gingival inflammation, pain, pocket formation, gingival withdrawal, increased bleeding and wound contamination occurred following retraction cord application. However, it is a known fact that the impression material is distorted or the accuracy of the measurement is decreased with the measurements taken without retraction. Nowadays, CAD / CAM (computer-aided design / computer-aided manufacturing) devices, which are designed to overcome these problems and eliminate the errors related to the measurement material, are the first step to be taken with a clear measure.Gingival retraction is recommended to improve the success of scanners in all restorations performed at the gingival or subgingival endpoint. Therefore, in our study, crown restorations will be produced from hybrid blocks by means of CAD / CAM device in order to evaluate the interaction of gingival health with hybrid blocks and to provide the latest technology and standardization.

ELIGIBILITY:
Inclusion Criteria:

* Being systemically healthy
* To indicate crown restoration in mandibular molar teeth
* To be vital to the preparation of the crown of the teeth

Exclusion Criteria:

* Systemically unhealthy individuals
* Endodontic treatment of mandibular molar teeth
* Mandibular molar female individuals drawn for various reasons
* Pregnant women
* Periodontally unhealthy individuals

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2020-01-17 (Actual); Study Completion 2020-04-17 (Actual)

PRIMARY OUTCOMES:
Retraction methods or procedures effects on gingival health | 3-12 months
  Probing depth is one of the criteria that shows the gingival health. In each control sessions same researcher measure the probing depth as mm via a periodontal probe.

CONTACTS AND LOCATIONS:
Locations (1):
- Beyza Ünalan Değirmenci, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Padbury A Jr, Eber R, Wang HL. Interactions between the gingiva and the margin of restorations. J Clin Periodontol. 2003 May;30(5):379-85. doi: 10.1034/j.1600-051x.2003.01277.x. PMID 12716328
- [Result] Al-Ani A, Bennani V, Chandler NP, Lyons KM, Thomson WM. New Zealand dentists' use of gingival retraction techniques for fixed prosthodontics and implants. N Z Dent J. 2010 Sep;106(3):92-6. PMID 20882737
- [Result] Goldberg PV, Higginbottom FL, Wilson TG. Periodontal considerations in restorative and implant therapy. Periodontol 2000. 2001;25:100-9. doi: 10.1034/j.1600-0757.2001.22250108.x. PMID 11155185
- [Result] Kopac I, Cvetko E, Marion L. Gingival inflammatory response induced by chemical retraction agents in beagle dogs. Int J Prosthodont. 2002 Jan-Feb;15(1):14-9. PMID 11887594
- [Result] Polat NT, Ozdemir AK, Turgut M. Effects of gingival retraction materials on gingival blood flow. Int J Prosthodont. 2007 Jan-Feb;20(1):57-62. PMID 17319365
- [Result] Ferrari M, Cagidiaco MC, Ercoli C. Tissue management with a new gingival retraction material: a preliminary clinical report. J Prosthet Dent. 1996 Mar;75(3):242-7. doi: 10.1016/s0022-3913(96)90479-5. PMID 8648569
- [Result] de Gennaro GG, Landesman HM, Calhoun JE, Martinoff JT. A comparison of gingival inflammation related to retraction cords. J Prosthet Dent. 1982 Apr;47(4):384-6. doi: 10.1016/s0022-3913(82)80085-1. PMID 6951037
- [Result] Ahmed SN, Donovan TE. Gingival displacement: Survey results of dentists' practice procedures. J Prosthet Dent. 2015 Jul;114(1):81-5.e1-2. doi: 10.1016/j.prosdent.2014.11.015. Epub 2015 Apr 24. PMID 25917854